CLINICAL TRIAL: NCT00293787
Title: A Study of Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-03
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle; glaucoma; ocular; hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — Travoprost; Timolol; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Travoprost 0.004%/Timolol 0.5% (Experimental): Travoprost 0.004%/Timolol 0.5% in both eyes each morning at 8 a.m. and Timolol vehicle in both eyes each evening at 8 p.m. for 3 months
  Interventions: Drug: Travoprost 0.004% / Timolol 0.5% Ophthalmic Solution; Other: Timolol Vehicle
- Xalatan + Timolol 0.5% (Active Comparator): Timolol 0.5% in both eyes each morning at 8 a.m. and Xalatan in both eyes each evening at 8 p.m. for 3 months
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution (XALATAN); Drug: Timolol Maleate Ophthalmic Solution 0.5%

INTERVENTIONS:
Drug: Travoprost 0.004% / Timolol 0.5% Ophthalmic Solution — Investigational ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: Travoprost 0.004%/Timolol 0.5%
Other: Timolol Vehicle — Placebo
  Arms: Travoprost 0.004%/Timolol 0.5%
Drug: Latanoprost 0.005% Ophthalmic Solution (XALATAN) — Commercially marketed ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension
  Other Names: XALATAN
  Arms: Xalatan + Timolol 0.5%
Drug: Timolol Maleate Ophthalmic Solution 0.5% — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension
  Arms: Xalatan + Timolol 0.5%

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of an investigational therapy for treating patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Diagnosis of open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component) or ocular hypertension.
* Mean IOP in each eye less than 18 mmHg at the screening visit.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant.
* History of chronic or recurrent severe inflammatory eye disease.
* Ocular trauma within the past six months in either eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Mean intraocular pressure (IOP) change at 3 months from baseline | 3 months